CLINICAL TRIAL: NCT02072850
Title: Cardiac Magnetic Resonance Imaging: New Pathological Insights and Their Functional and Clinical Significance in ST Elevation Acute Myocardial Infarction.
Brief Title: Detection and Significance of Heart Injury in ST Elevation Myocardial Infarction.
Acronym: BHF MR-MI
Status: Active, not recruiting | Type: Observational
Sponsor: NHS National Waiting Times Centre Board (Other)
Collaborators: Siemens Healthcare Diagnostics Inc (Industry); British Heart Foundation (Other)
Responsible Party: Principal Investigator, Colin Berry, Professor of Cardiology and Imaging, University of Glasgow
Other Study IDs: 10/S0703/28; Research grant number (Other Grant/Funding Number: British Heart Foundation PG/11/2/28474); Government health research (Other Grant/Funding Number: National Institute of Health Research (NIHR) Portfolio 10601)
Record Dates: First submitted 2014-02-25; First posted 2014-02-27 (Estimated); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Acute ST-elevation Myocardial Infarction
Keywords: Myocardial infarction; Primary percutaneous coronary intervention (PCI); Thrombolysis; Rescue PCI; Electrocardiogram; Magnetic resonance imaging; Area-at-risk; Myocardial salvage; Infarct size; Pressure wire; Coronary thermodilution; Coronary microvascular function; Index of microvascular resistance; Heart failure; Prognosis
MeSH Terms: conditions — Myocardial Infarction; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and urine samples have been archived.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Myocardial infarction: Patients presenting with acute-ST elevation myocardial infarction referred for emergency invasive management by primary or rescue percutaneous coronary intervention.
  Interventions: Device: Coronary pressure wire; Other: Magnetic resonance imaging of the heart

INTERVENTIONS:
Device: Coronary pressure wire — Guidewire-based coronary pressure- and temperature recordings (coronary thermodilution) with and without hyperaemia induced by intravenous administration of adenosine (140 ug/kg/min) in patients with acute ST-elevation myocardial infarction treated by emergency PCI.
  Other Names: Pressure wire Certus (St Jude Medical)
Other: Magnetic resonance imaging of the heart — Cardiac magnetic resonance imaging (MRI) with gadolinium contrast imaging at baseline (~ day 2) and 6 months (all participants) and in 30 subjects at 4 time-points (< 12 hours, days 2, 7-10 and at 6 months).
  Other Names: Cardiac MRI

SUMMARY:
Heart imaging with magnetic resonance imaging (MRI) provides detailed insights into heart function and injury. The nature and significance of heart injury after a heart attack is incompletely understood. We propose a 'natural history' study of heart attack injury using contemporary MRI methods. In a large hospital in the West of Scotland, heart attack patients will be invited to have at least two MRI scans and also continue with life-long follow-up. The results from the MRI scans will be assessed with all of the other clinical information obtained at the time of the heart attack and during follow-up. The results of our study should provide new insights into heart attack injury and these results should help improve how heart attack patients should be treated.

DETAILED DESCRIPTION:
Magnetic resonance imaging (MRI) provides detailed insights into soft tissue characteristics and this technique has particular value for imaging patients with acute myocardial infarction (MI). Recent advances in MRI have the potential to reveal new insights into the evolution and functional significance of myocardial injury and repair.

Here, we will study at least 300 consecutive patients with acute ST elevation MI (STEMI) and focus on oedema, scar and bleeding in the heart using MRI in patients managed by emergency percutaneous coronary intervention (PCI). Cardiac MRI scans will be performed at 1.5 Tesla (MAGNETOM, Siemens Healthcare). MRI will be used to assess initial heart function and injury. Myocardial salvage and haemorrhage are prioritised outcomes. Novel MRI methods will also be used to quantify the extent of myocardial jeopardy representing the initial area-at-risk (AAR), and the nature of this injury (strain, haemorrhage). The MRI methods will include T1, T2 and T2* relaxometry (mapping). Secondly, we will assess coronary artery disease severity by angiography and coronary artery function at the time of the heart attack treatment using a pressure-sensitive coronary guidewire (St Jude Medical). This wire can be used instead of the usual coronary wire and can provide information on heart injury, which can be linked in turn to the MRI findings. All of this information will be linked with health outcomes in the longer term.

We hypothesise that myocardial salvage, oedema, haemorrhage, and strain as revealed by MRI, have functional and prognostic significance. In all patients MRI will be performed at baseline (~day 2) and again at 6 months. In a subgroup of 30 patients, MRI will be performed on days <12 hours, and days 2, 7-10 days and 6 months post-MI. A blood and urine sample and quality of life will be obtained at baseline and at 6 months post-MI. Clinical outcomes (e.g. rehospitalisation, death) will be assessed at the end of the study (minimum 1 year) and again during longer term follow-up (minimum 3 years, maximum 20 years) by electronic linkage through central National Health Service (NHS) and government health records in order to determine the long-term prognostic significance of our initial observations with angiography, MRI and the pressure wire. The main statistical analyses will be conducted by an independent trials unit statistician.

ELIGIBILITY:
Inclusion Criteria:

* Acute STEMI

Exclusion Criteria:

* Major systemic illness (e.g. cancer limiting survival < 6 months);
* Metallic implant (e.g. cochlear implant);
* Metallic foreign body
* Pregnancy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a diagnosis of ST-elevation myocardial infarction (STEMI).
Sampling Method: Non-Probability Sample
Enrollment: 324 (Actual)
Dates: Start 2011-05 (Actual); Primary Completion 2012-11 (Actual); Study Completion 2031-05-01 (Estimated)

PRIMARY OUTCOMES:
Myocardial salvage | Baseline and 6 months after date of index hospitalisation for STEMI
  Myocardial salvage (% left ventricular volume) was defined as the difference between the initial jeopardised area-at-risk revealed by T2-weighted MRI (1.5 Tesla, Siemens Healthcare) at baseline and final infarct size revealed by contrast-enhanced MRI at 6 months on the same MRI scanner.

SECONDARY OUTCOMES:
Myocardial salvage index | Baseline and 6 months
  The myocardial salvage index was defined as infarct size at 6 months indexed to the initial area-at-risk revealed by T2-weighted MRI.
Final infarct size | MRI scan at 6 months after index hospitalisation
  Final infarct size imaged on the MRI scan 6 months after initial hospitalisation for STEMI. Late gadolinium enhancement is revealed by MRI scanning 10 - 15 minutes after intravenous gadolinium contrast administration. The myocardial mass of late gadolinium (grams) will be quantified by a semi-automatic detection method using a signal intensity threshold of >5 standard deviations above a remote reference region.
Myocardial haemorrhage | Baseline MRI scan
  Myocardial haemorrhage (a prioritised secondary outcome) is revealed by T2 weighted imaging and is defined as a confluent dark zone with a mean signal intensity <2 standard deviations of the mean signal intensity of the surrounding affected brighter area in the area of injury. Haemorrhage is specifically identified by T2* mapping, and will also be imaged with T2-weighted MRI (e.g. T2 mapping).
Microvascular obstruction | Baseline MRI scan
  MVO is classified as present (central dark zone with a subendocardial or intra-mural distribution (binary)) and non-relevant (dots or nil) and quantified as a % of total left ventricular mass, after adjustment for the initial area-at-risk revealed by T2-weighted MRI. Late MVO is imaged by MRI 10 - 15 minutes after contrast administration. Late MVO should be preceded by abnormal first pass and early MVO on 1, 3, and 5 minute scans.
First pass MVO | Baseline MRI
  First pass MVO is revealed by MRI scanning during the 'first pass' of gadolinium contrast in the ventricular myocardium. The extent of the first pass perfusion deficit at rest (i.e. first pass 'wash-in' MVO) will be assessed.
Early MVO | Baseline MRI
  Early MVO is acquired with MRI scanning 1 minute after gadolinium administration and forms part of the diagnostic criteria to confirm LATE MVO.
Area-at-risk | Baseline MRI scan
  The jeopardised area-at-risk on each axial image is defined as the percentage of left ventricular area delineated by the hyperintense zone on T2-weighted MRI with parametric maps. The initial area-at-risk will be assessed retrospectively with MRI ~2 days after initial hospitalisation for STEMI. Area-at-risk will be assessed with T2 and T1 mapping. The area-at-risk will be quantified by a semi-automatic detection method using a signal intensity threshold of >2 standard deviations above a remote reference region.
Myocardial T1 time | Baseline and follow-up MRI at 6 months
  The myocardial T1 relaxation time (ms) pre- and post-contrast will be estimated using a Modified Look-Locker Inversion recovery method (MOLLI, Siemens Healthcare). Post-contrast MOLLI scans will be obtained approximately 15 minutes after intravenous injection of gadolinium. Haematocrit will be measured from a full blood count blood test obtained at the time of the scan.
Myocardial T2 time | Baseline and follow-up MRI at 6 months
  The myocardial T2 relaxation time (ms) will be estimated using a balanced steady state free precession method (Siemens Healthcare).
Left ventricular ejection fraction | Baseline and follow-up MRI at 6 months
  Left ventricular ejection fraction (LVEF) is measured by subtraction of left ventricular end-systolic volume from left ventricular end-diastolic volume. LVEF is measure of systolic function and is a prognostically validated surrogate of health outcome.
Left ventricular end-diastolic volume | Baseline and follow-up MRI at 6 months
  Left ventricular end-diastolic volume (millilitres)
Left ventricular end-systolic volume | Baseline and follow-up MRI at 6 months
  Left ventricular end-systolic volume (millilitres)
Index of microvascular resistance | Day 0 at initial hospital admission
  The index of microvascular resistance (IMR) is a guidewire-derived measurement of coronary microvascular function. IMR = mean distal coronary pressure x mean transit time, measured during systemic hyperaemia induced by intravenous adenosine (140 ug/kg/min). Resting physiological parameters will also be measured.
Quality of life | Baseline and 6 months
  Patient-reported quality of life and health status will be assessed at baseline and during follow-up at 6 months. The Euroquol EQ-5D questionnaire will be used. Health-related quality of life will be related to other clinical information, including the MRI findings, and for estimation of quality-adjusted life years which is relevant for health economic assessments.
Recurrent myocardial infarction | 6 months
  The clinical characteristics that might predict recurrent cardiac events in survivors of STEMI are uncertain. The risk of recurrent MI is clinically relevant since this risk is potentially modifiable by additional PCI, as observed in the Preventative Angioplasty in Acute Myocardial Infarction (PRAMI) trial (N Engl J Med 2013 DOI: 10.1056/NEJMoa1305520).
  The clinical predictors of recurrent MI, as revealed by contrast MRI at 6 months and recurrent adverse cardiac events during the longer term will be assessed. Recurrent MI may be fatal or non-fatal. The characteristics to be assessed at baseline will include clinical characteristics (e.g. age, diabetes), coronary artery disease characteristics (as revealed by quantitative coronary analysis and plaque characterisation), guidewire-derived parameters of coronary artery function, and MI characteristics as revealed by contrast-enhanced MRI.
Adenosine response | Baseline
  The response to intravenous adenosine as reflected by patient-reported symptoms and changes in heart rate and blood pressure will be prospectively assessed. Adverse events, such as abnormalities in heart rate and rhythm and bronchospasm, that might be associated with the adenosine infusion will also be recorded.
MACE | Minimum 12 months
  Major Adverse Cardiac Events are defined as cardiac death, non-fatal myocardial infarction (MI) or hospitalisation for heart failure. The event definitions will follow the FDA guidelines (Hicks K et al 2010, 2012) and the Third Universal Definition of Myocardial Infarction (Thygesen et al Eur Heart J 2012). Events will be reviewed by a cardiologist who is independent of the research team and who is blinded to the MRI results. MACE will be related to the clinical and MRI findings at baseline. The survival analysis will be performed at the end of the study and again after a minimum of 3 years follow-up in all participants. The longer term follow-up will be performed by electronic case record linkage to hospital, NHS and government records.
MACCE | Minimum 12 months
  Major Adverse Cardiovascular Events (MACCE) is the composite of cardiovascular death, non-fatal MI, hospitalisation for TIA or stroke. The event definitions will follow the FDA guidelines (Hicks K et al 2010, 2012) and the Third Universal Definition of Myocardial Infarction (Thygesen et al Eur Heart J 2012). THE MACCE events will be reviewed by a cardiologist who is independent of the research team and who is blinded to the MRI results. MACCE will be related to the clinical and MRI findings at baseline. The survival analysis will be performed at the end of the study and again after a minimum of 3 years follow-up in all participants. The longer term follow-up will be performed by electronic case record linkage to hospital, NHS and government records.
Serious adverse cardiovascular events. | Minimum 12 months
  All serious adverse cardiovascular events including cardiovascular death, non-fatal MI, hospitalisation for unstable angina, hospitalisation for heart failure, implantable defibrillator implantation, hospitalisation for TIA or stroke, PCI, or CABG will be evaluated. Event definitions will follow the FDA guideline (Hicks K et al 2010, 2012) and the Third Universal Definition of Myocardial Infarction (Thygesen et al Eur Heart J 2012). In order to understand the prognostic significance of the clinical and MRI findings, these baseline findings will be associated with the cardiovascular events. The events will be reviewed by a cardiologist who is independent of the research team and who is blinded to the MRI results. The follow-up analysis will be performed at the end of the study and again after a min 3 years follow-up. The longer term follow-up will be performed by electronic case record linkage to hospital, NHS and government records.
All-cause death or heart failure | Minimum 12 months from baseline
  All-cause death and hospitalisation for heart failure is taken to be prognostically important and mechanistically linked to impaired heart function and injury after STEM. Event definitions will follow the FDA guideline (Hicks K et al 2010, 2012). In order to understand the prognostic significance of the clinical and MRI findings, these baseline findings will be associated with the occurrence of death or heart failure. Implantation of a cardiac defibrillator for primary or secondary prevention in a post-MI patient will also be considered. The events will be reviewed by a cardiologist who is independent of the research team and who is blinded to the MRI results. The follow-up analysis will be performed at the end of the study and again after a minimum of 3 years follow-up in all participants. The longer term follow-up will be performed by electronic case record linkage to hospital, NHS and government records.

CONTACTS AND LOCATIONS:
Overall Officials: Colin Berry, MB ChB BSc PhD FRCP FACC, Principal Investigator — University of Glasgow
Locations (1):
- Golden Jubilee National Hospital, Clydebank, Dunbartonshire, United Kingdom

REFERENCES:
- [Background] Ahmed N, Layland J, Carrick D, Petrie MC, McEntegart M, Eteiba H, Hood S, Lindsay M, Watkins S, Davie A, Mahrous A, Carberry J, Teng V, McConnachie A, Curzen N, Oldroyd KG, Berry C. Safety of guidewire-based measurement of fractional flow reserve and the index of microvascular resistance using intravenous adenosine in patients with acute or recent myocardial infarction. Int J Cardiol. 2016 Jan 1;202:305-10. doi: 10.1016/j.ijcard.2015.09.014. Epub 2015 Sep 18. PMID 26418191
- [Background] Carberry J, Carrick D, Haig C, Ahmed N, Mordi I, McEntegart M, Petrie MC, Eteiba H, Hood S, Watkins S, Lindsay M, Davie A, Mahrous A, Ford I, Sattar N, Welsh P, Radjenovic A, Oldroyd KG, Berry C. Persistent Iron Within the Infarct Core After ST-Segment Elevation Myocardial Infarction: Implications for Left Ventricular Remodeling and Health Outcomes. JACC Cardiovasc Imaging. 2018 Sep;11(9):1248-1256. doi: 10.1016/j.jcmg.2017.08.027. Epub 2017 Nov 15. PMID 29153575
- [Background] Bulluck H, Carberry J, Carrick D, McEntegart M, Petrie MC, Eteiba H, Hood S, Watkins S, Lindsay M, Mahrous A, Ford I, Oldroyd KG, Berry C. Redefining Adverse and Reverse Left Ventricular Remodeling by Cardiovascular Magnetic Resonance Following ST-Segment-Elevation Myocardial Infarction and Their Implications on Long-Term Prognosis. Circ Cardiovasc Imaging. 2020 Jul;13(7):e009937. doi: 10.1161/CIRCIMAGING.119.009937. Epub 2020 Jul 21. PMID 32689822
- [Background] Carberry J, Carrick D, Haig C, Rauhalammi SM, Ahmed N, Mordi I, McEntegart M, Petrie MC, Eteiba H, Hood S, Watkins S, Lindsay M, Davie A, Mahrous A, Ford I, Sattar N, Welsh P, Radjenovic A, Oldroyd KG, Berry C. Remote Zone Extracellular Volume and Left Ventricular Remodeling in Survivors of ST-Elevation Myocardial Infarction. Hypertension. 2016 Aug;68(2):385-91. doi: 10.1161/HYPERTENSIONAHA.116.07222. Epub 2016 Jun 27. PMID 27354423
- [Background] Yew SN, Carrick D, Corcoran D, Ahmed N, Carberry J, Teng Yue May V, McEntegart M, Petrie MC, Eteiba H, Lindsay M, Hood S, Watkins S, Davie A, Mahrous A, Mordi I, Ford I, Oldroyd KG, Berry C. Coronary Thermodilution Waveforms After Acute Reperfused ST-Segment-Elevation Myocardial Infarction: Relation to Microvascular Obstruction and Prognosis. J Am Heart Assoc. 2018 Aug 7;7(15):e008957. doi: 10.1161/JAHA.118.008957. PMID 30371237
- [Background] Carrick D, Haig C, Carberry J, May VTY, McCartney P, Welsh P, Ahmed N, McEntegart M, Petrie MC, Eteiba H, Lindsay M, Hood S, Watkins S, Mahrous A, Rauhalammi SM, Mordi I, Ford I, Radjenovic A, Sattar N, Oldroyd KG, Berry C. Microvascular resistance of the culprit coronary artery in acute ST-elevation myocardial infarction. JCI Insight. 2016 May 5;1(6):e85768. doi: 10.1172/jci.insight.85768. PMID 27699259
- [Background] Mangion K, Carrick D, Carberry J, Mahrous A, McComb C, Oldroyd KG, Eteiba H, Lindsay M, McEntegart M, Hood S, Petrie MC, Watkins S, Davie A, Zhong X, Epstein FH, Haig CE, Berry C. Circumferential Strain Predicts Major Adverse Cardiovascular Events Following an Acute ST-Segment-Elevation Myocardial Infarction. Radiology. 2019 Feb;290(2):329-337. doi: 10.1148/radiol.2018181253. Epub 2018 Nov 20. PMID 30457480
- [Background] Haig C, Carrick D, Carberry J, Mangion K, Maznyczka A, Wetherall K, McEntegart M, Petrie MC, Eteiba H, Lindsay M, Hood S, Watkins S, Davie A, Mahrous A, Mordi I, Ahmed N, Teng Yue May V, Ford I, Radjenovic A, Welsh P, Sattar N, Oldroyd KG, Berry C. Current Smoking and Prognosis After Acute ST-Segment Elevation Myocardial Infarction: New Pathophysiological Insights. JACC Cardiovasc Imaging. 2019 Jun;12(6):993-1003. doi: 10.1016/j.jcmg.2018.05.022. Epub 2018 Jul 18. PMID 30031700
- [Background] Maznyczka AM, Carrick D, Carberry J, Mangion K, McEntegart M, Petrie MC, Eteiba H, Lindsay M, Hood S, Watkins S, Davie A, Mahrous A, Ford I, Welsh P, Sattar N, Oldroyd KG, Berry C. Sex-based associations with microvascular injury and outcomes after ST-segment elevation myocardial infarction. Open Heart. 2019 Apr 29;6(1):e000979. doi: 10.1136/openhrt-2018-000979. eCollection 2019. PMID 31168381
- [Background] Ahmed N, Carberry J, Teng V, Carrick D, Berry C. Risk assessment in patients with an acute ST-elevation myocardial infarction. J Comp Eff Res. 2016 Nov;5(6):581-593. doi: 10.2217/cer-2016-0017. Epub 2016 Sep 1. PMID 27580675
- [Background] Carrick D, Haig C, Maznyczka AM, Carberry J, Mangion K, Ahmed N, Yue May VT, McEntegart M, Petrie MC, Eteiba H, Lindsay M, Hood S, Watkins S, Davie A, Mahrous A, Mordi I, Ford I, Radjenovic A, Welsh P, Sattar N, Wetherall K, Oldroyd KG, Berry C. Hypertension, Microvascular Pathology, and Prognosis After an Acute Myocardial Infarction. Hypertension. 2018 Sep;72(3):720-730. doi: 10.1161/HYPERTENSIONAHA.117.10786. PMID 30012869
- [Background] Bulluck H, Carberry J, Carrick D, McCartney PJ, Maznyczka AM, Greenwood JP, Maredia N, Chowdhary S, Gershlick AH, Appleby C, Cotton JM, Wragg A, Curzen N, McEntegart M, Petrie MC, Eteiba H, Watkins S, Lindsay M, Mahrous A, Oldroyd KG, Berry C. A Noncontrast CMR Risk Score for Long-Term Risk Stratification in Reperfused ST-Segment Elevation Myocardial Infarction. JACC Cardiovasc Imaging. 2022 Mar;15(3):431-440. doi: 10.1016/j.jcmg.2021.08.006. Epub 2022 Jan 12. PMID 35272808
- [Background] Reindl M, Stiermaier T, Lechner I, Tiller C, Holzknecht M, Fink P, Mayr A, Klug G, Feistritzer HJ, Delewi R, Hirsch A, Carberry J, Carrick D, Bauer A, Metzler B, Nijveldt R, Thiele H, Berry C, Eitel I, Reinstadler SJ. Infarct severity and outcomes in ST-elevation myocardial infarction patients without standard modifiable risk factors - A multicenter cardiac magnetic resonance study. Eur J Intern Med. 2024 Jan;119:78-83. doi: 10.1016/j.ejim.2023.08.013. Epub 2023 Aug 25. PMID 37634958
- [Background] Lechner I, Reindl M, Stiermaier T, Tiller C, Holzknecht M, Oberhollenzer F, von der Emde S, Mayr A, Feistritzer HJ, Carberry J, Carrick D, Bauer A, Thiele H, Berry C, Eitel I, Metzler B, Reinstadler SJ. Clinical Outcomes Associated With Various Microvascular Injury Patterns Identified by CMR After STEMI. J Am Coll Cardiol. 2024 May 28;83(21):2052-2062. doi: 10.1016/j.jacc.2024.03.408. PMID 38777509
- [Background] El Farissi M, Zimmermann FM, De Maria GL, van Royen N, van Leeuwen MAH, Carrick D, Carberry J, Wijnbergen IF, Konijnenberg LSF, Hoole SP, Marin F, Fineschi M, Pijls NHJ, Oldroyd KG, Banning AP, Berry C, Fearon WF. The Index of Microcirculatory Resistance After Primary PCI: A Pooled Analysis of Individual Patient Data. JACC Cardiovasc Interv. 2023 Oct 9;16(19):2383-2392. doi: 10.1016/j.jcin.2023.08.030. PMID 37821183
- [Background] Carrick D, Haig C, Ahmed N, Carberry J, Yue May VT, McEntegart M, Petrie MC, Eteiba H, Lindsay M, Hood S, Watkins S, Davie A, Mahrous A, Mordi I, Ford I, Radjenovic A, Oldroyd KG, Berry C. Comparative Prognostic Utility of Indexes of Microvascular Function Alone or in Combination in Patients With an Acute ST-Segment-Elevation Myocardial Infarction. Circulation. 2016 Dec 6;134(23):1833-1847. doi: 10.1161/CIRCULATIONAHA.116.022603. Epub 2016 Nov 1. PMID 27803036
- [Background] Berry C, Carrick D, Haig C, Oldroyd KG. "Waves of Edema" Seem Implausible. J Am Coll Cardiol. 2016 Apr 19;67(15):1868-1869. doi: 10.1016/j.jacc.2015.11.073. No abstract available. PMID 27081030
- [Background] Mangion K, Corcoran D, Carrick D, Berry C. New perspectives on the role of cardiac magnetic resonance imaging to evaluate myocardial salvage and myocardial hemorrhage after acute reperfused ST-elevation myocardial infarction. Expert Rev Cardiovasc Ther. 2016 Jul;14(7):843-54. doi: 10.1586/14779072.2016.1173544. Epub 2016 Apr 26. PMID 27043975
- [Background] Carrick D, Haig C, Ahmed N, Rauhalammi S, Clerfond G, Carberry J, Mordi I, McEntegart M, Petrie MC, Eteiba H, Hood S, Watkins S, Lindsay MM, Mahrous A, Welsh P, Sattar N, Ford I, Oldroyd KG, Radjenovic A, Berry C. Temporal Evolution of Myocardial Hemorrhage and Edema in Patients After Acute ST-Segment Elevation Myocardial Infarction: Pathophysiological Insights and Clinical Implications. J Am Heart Assoc. 2016 Feb 23;5(2):e002834. doi: 10.1161/JAHA.115.002834. PMID 26908408
- [Background] Carrick D, Haig C, Ahmed N, McEntegart M, Petrie MC, Eteiba H, Hood S, Watkins S, Lindsay MM, Davie A, Mahrous A, Mordi I, Rauhalammi S, Sattar N, Welsh P, Radjenovic A, Ford I, Oldroyd KG, Berry C. Myocardial Hemorrhage After Acute Reperfused ST-Segment-Elevation Myocardial Infarction: Relation to Microvascular Obstruction and Prognostic Significance. Circ Cardiovasc Imaging. 2016 Jan;9(1):e004148. doi: 10.1161/CIRCIMAGING.115.004148. PMID 26763281
- [Background] Carrick D, Haig C, Rauhalammi S, Ahmed N, Mordi I, McEntegart M, Petrie MC, Eteiba H, Hood S, Watkins S, Lindsay M, Mahrous A, Ford I, Tzemos N, Sattar N, Welsh P, Radjenovic A, Oldroyd KG, Berry C. Prognostic significance of infarct core pathology revealed by quantitative non-contrast in comparison with contrast cardiac magnetic resonance imaging in reperfused ST-elevation myocardial infarction survivors. Eur Heart J. 2016 Apr 1;37(13):1044-59. doi: 10.1093/eurheartj/ehv372. Epub 2015 Aug 10. PMID 26261290
- [Background] Carrick D, Haig C, Rauhalammi S, Ahmed N, Mordi I, McEntegart M, Petrie MC, Eteiba H, Lindsay M, Watkins S, Hood S, Davie A, Mahrous A, Sattar N, Welsh P, Tzemos N, Radjenovic A, Ford I, Oldroyd KG, Berry C. Pathophysiology of LV Remodeling in Survivors of STEMI: Inflammation, Remote Myocardium, and Prognosis. JACC Cardiovasc Imaging. 2015 Jul;8(7):779-89. doi: 10.1016/j.jcmg.2015.03.007. Epub 2015 Jun 17. PMID 26093923
- [Background] Gao H, Carrick D, Berry C, Griffith BE, Luo X. Dynamic finite-strain modelling of the human left ventricle in health and disease using an immersed boundary-finite element method. IMA J Appl Math. 2014 Oct;79(5):978-1010. doi: 10.1093/imamat/hxu029. Epub 2014 Jul 1. PMID 27041786
- [Background] Layland J, Carrick D, Lee M, Oldroyd K, Berry C. Adenosine: physiology, pharmacology, and clinical applications. JACC Cardiovasc Interv. 2014 Jun;7(6):581-91. doi: 10.1016/j.jcin.2014.02.009. Epub 2014 May 14. PMID 24835328
- [Background] Carrick D, Oldroyd KG, McEntegart M, Haig C, Petrie MC, Eteiba H, Hood S, Owens C, Watkins S, Layland J, Lindsay M, Peat E, Rae A, Behan M, Sood A, Hillis WS, Mordi I, Mahrous A, Ahmed N, Wilson R, Lasalle L, Genereux P, Ford I, Berry C. A randomized trial of deferred stenting versus immediate stenting to prevent no- or slow-reflow in acute ST-segment elevation myocardial infarction (DEFER-STEMI). J Am Coll Cardiol. 2014 May 27;63(20):2088-2098. doi: 10.1016/j.jacc.2014.02.530. Epub 2014 Feb 27. PMID 24583294
- [Background] Ahmed N, Carrick D, Layland J, Oldroyd KG, Berry C. The role of cardiac magnetic resonance imaging (MRI) in acute myocardial infarction (AMI). Heart Lung Circ. 2013 Apr;22(4):243-55. doi: 10.1016/j.hlc.2012.11.016. Epub 2012 Dec 29. PMID 23279917
- [Background] Carrick D, Berry C. Prognostic importance of myocardial infarct characteristics. Eur Heart J Cardiovasc Imaging. 2013 Apr;14(4):313-5. doi: 10.1093/ehjci/jes296. Epub 2012 Dec 17. No abstract available. PMID 23248208
- [Background] Berry C, McEntegart M, Petrie MC, Eteiba H, Lindsay M, Hood S, Watkins S, Davie A, Carrick D, Payne AR, McGeoch RJ, Oldroyd KG. Meta-Analysis of the Index of Microvascular Resistance in Acute STEMI Using Incomplete Data. JACC Cardiovasc Interv. 2017 Feb 27;10(4):421-422. doi: 10.1016/j.jcin.2016.12.268. No abstract available. PMID 28231914
- [Background] Gao H, Mangion K, Carrick D, Husmeier D, Luo X, Berry C. Estimating prognosis in patients with acute myocardial infarction using personalized computational heart models. Sci Rep. 2017 Oct 19;7(1):13527. doi: 10.1038/s41598-017-13635-2. PMID 29051544
- [Background] Carberry J, Carrick D, Haig C, Ahmed N, Mordi I, McEntegart M, Petrie MC, Eteiba H, Hood S, Watkins S, Lindsay M, Davie A, Mahrous A, Ford I, Sattar N, Welsh P, Radjenovic A, Oldroyd KG, Berry C. Persistence of Infarct Zone T2 Hyperintensity at 6 Months After Acute ST-Segment-Elevation Myocardial Infarction: Incidence, Pathophysiology, and Prognostic Implications. Circ Cardiovasc Imaging. 2017 Dec;10(12):e006586. doi: 10.1161/CIRCIMAGING.117.006586. PMID 29242240
- [Background] Mangion K, Carrick D, Clerfond G, Rush C, McComb C, Oldroyd KG, Petrie MC, Eteiba H, Lindsay M, McEntegart M, Hood S, Watkins S, Davie A, Auger DA, Zhong X, Epstein FH, Haig CE, Berry C. Predictors of segmental myocardial functional recovery in patients after an acute ST-Elevation myocardial infarction. Eur J Radiol. 2019 Mar;112:121-129. doi: 10.1016/j.ejrad.2019.01.010. Epub 2019 Jan 14. PMID 30777200
- [Background] Maznyczka AM, Carrick D, Oldroyd KG, James-Rae G, McCartney P, Greenwood JP, Good R, McEntegart M, Eteiba H, Lindsay MM, Cotton JM, Petrie MC, Berry C. Thermodilution-derived temperature recovery time: a novel predictor of microvascular reperfusion and prognosis after myocardial infarction. EuroIntervention. 2021 Jun 25;17(3):220-228. doi: 10.4244/EIJ-D-19-00904. PMID 32122822
- See also: Chief Scientist Office, NHS Scotland and Healthscience Scotland — http://www.nhsresearchscotland.org.uk/research-in-scotland
- See also: British Heart Foundation — https://www.bhf.org.uk/research